CLINICAL TRIAL: NCT00503204
Title: A Phase I, Open Label, Multi-Centre Study to Assess the Safety and Tolerability of Cediranib (RECENTIN™, AZD2171) in Combination With Lomustine Chemotherapy for Patients With Primary Recurrent Malignant Brain Tumours for Whom Lomustine Would be a Standard Therapy
Brief Title: Phase I : Cediranib in Combination With Lomustine Chemotherapy in Recurrent Malignant Brain Tumour
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jane Robertson, Medical Science Director, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00057; EuDract 2007-000909-30
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Recurrent Glioblastoma; Brain Tumor
Keywords: cancer; tumor; advance solid tumour; glioblastoma; malignant brain tumour
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Neoplasms | interventions — cediranib; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Lomustine + Cediranib (AZD2171)
  Interventions: Drug: Cediranib; Drug: Lomustine

INTERVENTIONS:
Drug: Cediranib — oral tablet
  Other Names: RECENTIN™; AZD2171
Drug: Lomustine — oral capsule
  Other Names: CCNU; CeeNU®

SUMMARY:
This is a Phase I, open-label, multi-centre study designed to assess the safety and tolerability of Cediranib in combination with lomustine in patients with primary recurrent malignant brain tumour.

ELIGIBILITY:
Inclusion Criteria:

* Primary recurrent malignant brain tumour for whom lomustine would be standard therapy - diagnosis & stage
* Patients received no more than 2 previous systemic chemotherapy regimes
* Life Expectancy > 12 weeks
* Patients must be at least 3 months from the completion of cranial radiation therapy

Exclusion Criteria:

* History of poorly controlled high blood pressure
* Recent major surgery prior to entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of cediranib in combination with oral lomustine and to confirm a dose for further studies with this combination. | Assessed at each visit

SECONDARY OUTCOMES:
Compare the pharmacokinetics of cediranib alone versus when in combination with lomustine as measured by minimum steady state plasma concentration (Css,min) steady-state plasma concentration | assessed 2 & 4 hours post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca; Tracy Batchelor, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Research Site, Boston, Massachusetts, United States
- Research Site, Sutton, United Kingdom